CLINICAL TRIAL: NCT06441383
Title: Assessment of Sleep Disordersin People Living With HIV in the Era of New Antiretroviral Therapies in North of France
Acronym: SANDMAN
Status: Not yet recruiting | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHT/URC/2023/11
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections; Sleep Disorder
MeSH Terms: conditions — HIV Infections; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pittsburgh Sleep Quality Index — The the Pittsburg Sleep Quality Index (PSQI) questionnaire is a standardized tool for the subjective assessment of sleep. Sleep is described according to 7 components: subjective sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disorders, medication use and daytime dysfunction. The sum of the scores for these 7 components gives an overall score of 21 points maximum.
  The presence of sleep disorders will be defined according to the results of the PSQI, with a value above 5 defining the presence of sleep disorders.

SUMMARY:
People living with HIV (PLHIV) appear to present with sleep-related complaints more frequently than the general population, with a prevalence of 50-70%. The latest French multi-center epidemiological data are dated. The prevalence of the different types of sleep disorders, however, is poorly documented, with the literature focusing mainly on insomnia and neuropsychological disorders that can lead to sleep disorder-like symptoms, and on the impact of antiretroviral drugs in particular. However, there are other sleep disorders such as sleep apnea syndrome (SAHOS) or restless legs syndrome. SAHOS has been studied in small series of patients.

This multicenter, cross-sectional study will identify and update the functional complaints presented by PLHIV, estimate the prevalence of people at high risk of sleep apnea syndrome, and study the associated socio-demographic factors, in relation to HIV infection and antiretrovirals. This study could open up avenues for new management approaches and earlier detection of sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* PLHIV usually treated at referral centers in northern France.

Exclusion Criteria:

* Minor patient;
* Patient with insufficient understanding of the French language, as judged by the investigator;
* Patient unable to give free and informed consent;
* Refusal to participate;
* Patient under legal protection, guardianship or curatorship;
* Pregnant and breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is all adults living with HIV. The study will be offered to all PLHIV at the time of their annual specialist consultation with their infectiologist in the referring hospital centers in northern France.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disorders | at baseline
  The presence of sleep disorders will be defined according to the results of the Pittsburg Sleep Quality Index (PSQI), with a value greater than 5 defining the presence of sleep disorders.

SECONDARY OUTCOMES:
Prevalence of Obstructive Sleep Apnea-Hypopnea Syndrome | at baseline
  The Berlin score defines the signs suggestive of Obstructive Sleep Apnea-Hypopnea Syndrome. A score ≥ 2 positive categories will define a high risk of Obstructive Sleep Apnea-Hypopnea Syndrome
Prevalence of Restless Legs Syndrome | at baseline
  The International Restless Legs Syndrome (RLS) Severity Scale will identify patients with symptoms in favor of RLS.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No